CLINICAL TRIAL: NCT04339829
Title: An Open Label, Multicenter, Phase II Study of Dacomitinib for EGFR Mutated Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Lu shun, Vice-chairman, Guangdong Association of Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2001
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Dacomitinib for EGFR Mutated Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Intervention Model Description: This is a multi-center, single-arm, open-label, Phase 2 clinical study of Dacomitinib for EGFR Mutated Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dacomitinib 45mg PO ,QD (Other): Single arm
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Dacomitinib orally on a continuous daily basis at a starting dose of 45 mg QD

SUMMARY:
This is a multi-center, single-arm, open-label, Phase 2 clinical study of Dacomitinib for EGFR Mutated Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases.

DETAILED DESCRIPTION:
The brain is a common site of metastases among patients with non-small-cell lung cancer (NSCLC).The incidence of CNS metastases in patients with EGFR mutation-positive NSCLC is 24% at first diagnosis almost doubles over the course of the disease. Several data has shown treatment with first generation EGFR-tyrosine kinase inhibitors (TKIs) can reduce the risk of progression in the CNS, compared with chemotherapy or WBRT.Pre-clinical data showing that brain homogenate dacomitinib concentrations is similar to plasma in mice. While, there are evidence show that dacomitinib have efficacy in NSCLC patients with BM. This phase II study was designed to prospectively evaluate the efficacy and safety of Dacomitinib in NSCLC patients with BM.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a voluntarily given, personally signed and dated, written informed consent document;
* Age≥18 years, male or female;
* The presence of an EGFR activating mutation (exon 19 deletion or the L858R mutation in exon 21) in tumor specimen determined by the local laboratory. It is acceptable for subjects with the presence of the exon 20 T790M mutation together with either EGFR activating mutation (exon 19 deletion or the L858R mutation in exon 21) to be included in this study;
* Evidence of newly diagnosed stage IIIB/IV (based on Union for International Cancer Control (UICC) staging system version 7) or recurrent (minimum of 12 months disease free interval between completion of systemic therapy and recurrence of NSCLC required) NSCLC of adenocarcinoma histo- and/or cytopathology or its pathologically accepted variants using tumor specimen (assessed according to accepted standards by a local laboratory). For this purpose the World Health Organization/International Association of Study of Lung Cancer Histologic Classification of Lung Cancer Criteria will be used and the diagnosis of NSCLC NOS (not otherwise specified), squamous or mixed adeno-squamous lung carcinomas will not be allowed;
* Have an ECOG PS of 0 or 1;
* No prior treatment with systemic therapy for locally advanced or metastatic NSCLC. Completed neoadjuvant/adjuvant chemotherapy/immunotherapy and/or combined modality chemotherapy/radiation therapy permitted only in cases in which there is a minimum of 12 months disease free interval between completion of systemic therapy and recurrence of NSCLC. Prior treatment with an EGFR-TKI or other TKIs is not allowed;
* Brain metastases lesions should be more than or equal to 3 metastatic lesions in the brain . At least one target lesion's diameter among these lesions should be more than 1 centimeter（ Patients with CNS metastases. whose condition was neurologically stable were eligible. Any previous definitive treatment or glucocorticoid therapy had to be completed at least 2 weeks before initiation of the trial treatment.）.
* Radiologically measurable disease by RECIST v1.1 criteria:

  1. At least one target lesion that has not previously been radiated, and is measurable according to RECIST v1.1;
  2. Acceptable radiologic procedures for disease assessment include contrast enhanced conventional or spiral computed tomography (CT), or contrast enhanced magnetic resonance imaging (MRI); Non contrast CT scan is acceptable only for subjects who are both allergic to intravenous contrast and unable to cooperate with MRI, or MRI is not available. The following are not allowed as sole documentation of target lesions: CT component of positron emission tomography (PET)/CT, ultrasound alone, nuclear scans (including bone or PET scans), chest X-ray or bone radiographs, and tumor markers;
* Adequate organ function, including:

  1. Estimated creatinine clearance >30 mL/min (as determined by Cockcroft-Gault formula or the study site's standard formula);
  2. Urinary protein <3+ by urine dipstick. If urine protein by dipstick is ≥3+, then a urine protein/creatinine ratio (UPC) should be obtained. The subject may enter only if UPC is <2.0;
  3. Absolute neutrophil count (ANC) ≥1500 cells/mm3;
  4. Platelets ≥100,000 cells/mm3;
  5. Hemoglobin ≥10.0 g/dL；
  6. Bilirubin≤1.5 x ULN;
  7. AST (also known as SGOT) and ALT (also known as SGPT) <2.5 x ULN (<5.0 x ULN if hepatic metastases).
* Female subjects must be postmenopausal (defined as 12 months of amenorrhea following last menses), or they or their partners must be surgically sterile, or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the investigator using following criteria:

Acceptable contraception for women include implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence, or a partner who has been surgically sterile (e.g. by vasectomy) for at least 6 months. Acceptable contraception for a male includes surgical sterility (e.g. by vasectomy) for at least 6 months, sexual abstinence, or condoms plus spermicide.

* All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to starting study treatment;
* Male subjects or their female partners must be surgically sterile or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the investigator. Or female partners must be postmenopausal (defined as 12 months of amenorrhea following last menses);
* Willing and able to comply with study scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any evidence of mixed histo- and/or cytology that includes elements of small cell or carcinoid lung cancer. Variations of adenocarcinoma are allowed, however no squamous element can be present;
* Any other mutation other than exon 19 deletion or L858R in exon 21, with or without the presence of the exon 20 T790M mutation. Both mutations (exon 19 deletion and L858R mutation in exon 21) within a tumor sample;
* Symptomatic brain or leptomeningeal metastases, who are neurologically unstable or require increasing doses of steroids to manage CNS symptoms within two weeks prior to starting dacomitinib;
* Any previous anti-cancer systemic treatment of locally advanced, or metastatic NSCLC including but not limited to chemotherapy, targeted therapies, small molecules, EGFR-TKIs and other TKIs, monoclonal antibodies, anti-cancer vaccines, radiotherapy (other than palliative radiotherapy to lesions that will not be followed for tumor assessment on this study, i.e., non-target lesions). Completed neoadjuvant/adjuvant chemotherapy/immunotherapy and/or combined modality chemotherapy/ radiation therapy permitted only in cases in which there is a minimum of 12 months disease free interval between completion of systemic therapy and recurrence of NSCLC. Prior treatment with an EGFR-TKI or other TKIs is not allowed;
* Any surgery (not including minor procedures such as lymph node biopsy), palliative radiotherapy or pleurodesis within 2 weeks of baseline assessments;
* Any clinically significant gastrointestinal abnormalities that may impair intake, transit or absorption of the study drug, such as the inability to take oral medication;
* Current enrollment in another therapeutic clinical study;
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this study; or known drug abuse/alcohol abuse;
* History of, or currently suspected, diffuse non-infectious pneumonitis or interstitial lung disease including:

  1. Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease;
  2. Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline;
  3. Insufficient lung function as determined by either clinical examination or an arterial oxygen tension of <70 Torr.
* Any history of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Clinically important abnormalities in cardiac rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, second degree heart block, third degree heart block) OR:

  1. Diagnosed or suspected congenital long QT syndrome;
  2. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
  3. Prolonged QTc on ECG; QTc must be less than CTCAE v4.0 Grade 2 (≤480 msec) using Fridericia's or Bazett's correction formula with a manual reading by the investigator if required. The ECG may be repeated for evaluation of eligibility after management of correctable causes for observed QTc prolongation;
  4. Any history of second or third degree heart block;
  5. Heart rate <45 beats per minute on ECG in the presence of clinical symptoms (e.g., hypotension, evidence of hypoperfusion);
* Severely impaired (defined as Child-Pugh Class C) hepatic dysfunction;
* Prior malignancy: Subjects will not be eligible if they have history of, or evidence of active disease of another concurrent malignancy within the previous five years. Exception would be effectively treated past history of non melanoma skin cancer or in-situ cervical cancer with no evidence of active disease;
* Other severe acute or chronic medical condition that may increase the risk associated with study participation or investigational drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study;
* Use of narrow therapeutic index drugs that are CYP2D6 substrates (procainamide, pimozide, and thioridazine etc.) from screening to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival （PFS） | 20 months
  Progression Free Survival （PFS）is defined as the time from start of treatment to the date of disease progression as defined by RECIST v1.1 per investigator review or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Intracranial Objective Response Rate | 20 months
  Intracranial Objective Response Rate is defined as the proportion of subjects with a BOR of either CR or PR of intracranial disease, where BOR is the best response recorded from the start of treatment until disease progression or start of other anticancer therapy. As per RECIST v1.1 guidelines, PR and CR do not need to be confirmed following initial response documentation.
Objective Response Rate | 20 months
  Objective Response Rate is defined as the proportion of subjects with a BOR of either CR or PR, where BOR is the best response recorded from the start of treatment until disease progression or start of other anticancer therapy. As per RECIST v1.1 guidelines, PR and CR do not need to be confirmed following initial response documentation.
Disease control rate | 20 months
  Disease control rate is defined as the proportion of patients with complete response (CR) or partial response (PR) or subjects with stable disease (SD) as per investigator assessment according to RECIST 1.1 criteria.
Duration of response | 20 months
  Duration of response is defined as the time from first documented response of CR or PR to date of first documented progression or death due to any cause, according to RECIST 1.1 criteria
Intracranial Progression Free Survival | 20 months
  Intracranial Progression Free Survival is defined as confirmed by investigator with morphologically proven intracranial PD [presence of at least one key symptom in combination with radiologic evidence including CT or MRI of PD in the brain on follow-up or death due to any cause, whichever occurred first.
Overall Survival | 48 months
  Overall Survival is defined as the time from start of treatment to the date of death for any cause. In the absence of confirmation of death, survival time will be censored at the last date the subject is known to be alive.

REFERENCES:
- [Background] Gross ME, Shazer RL, Agus DB. Targeting the HER-kinase axis in cancer. Semin Oncol. 2004 Feb;31(1 Suppl 3):9-20. doi: 10.1053/j.seminoncol.2004.01.005. PMID 15052539
- [Background] Barnes CJ, Kumar R. Epidermal growth factor receptor family tyrosine kinases as signal integrators and therapeutic targets. Cancer Metastasis Rev. 2003 Dec;22(4):301-7. doi: 10.1023/a:1023726827771. PMID 12884907
- [Background] Arteaga C. Targeting HER1/EGFR: a molecular approach to cancer therapy. Semin Oncol. 2003 Jun;30(3 Suppl 7):3-14. PMID 12840796
- [Background] Baselga J, Hammond LA. HER-targeted tyrosine-kinase inhibitors. Oncology. 2002;63 Suppl 1:6-16. doi: 10.1159/000066198. PMID 12422050
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Roberts PJ, Stinchcombe TE, Der CJ, Socinski MA. Personalized medicine in non-small-cell lung cancer: is KRAS a useful marker in selecting patients for epidermal growth factor receptor-targeted therapy? J Clin Oncol. 2010 Nov 1;28(31):4769-77. doi: 10.1200/JCO.2009.27.4365. Epub 2010 Oct 4. PMID 20921461
- [Background] Ramalingam SS, Blackhall F, Krzakowski M, Barrios CH, Park K, Bover I, Seog Heo D, Rosell R, Talbot DC, Frank R, Letrent SP, Ruiz-Garcia A, Taylor I, Liang JQ, Campbell AK, O'Connell J, Boyer M. Randomized phase II study of dacomitinib (PF-00299804), an irreversible pan-human epidermal growth factor receptor inhibitor, versus erlotinib in patients with advanced non-small-cell lung cancer. J Clin Oncol. 2012 Sep 20;30(27):3337-44. doi: 10.1200/JCO.2011.40.9433. Epub 2012 Jul 2. PMID 22753918
- [Background] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Background] Mok TS, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Lee M, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Wu YL. Improvement in Overall Survival in a Randomized Study That Compared Dacomitinib With Gefitinib in Patients With Advanced Non-Small-Cell Lung Cancer and EGFR-Activating Mutations. J Clin Oncol. 2018 Aug 1;36(22):2244-2250. doi: 10.1200/JCO.2018.78.7994. Epub 2018 Jun 4. PMID 29864379
- [Background] Wu YL, Zhou C, Cheng Y, Lu S, Chen GY, Huang C, Huang YS, Yan HH, Ren S, Liu Y, Yang JJ. Erlotinib as second-line treatment in patients with advanced non-small-cell lung cancer and asymptomatic brain metastases: a phase II study (CTONG-0803). Ann Oncol. 2013 Apr;24(4):993-9. doi: 10.1093/annonc/mds529. Epub 2012 Nov 4. PMID 23129122
- [Background] Yang JJ, Zhou C, Huang Y, Feng J, Lu S, Song Y, Huang C, Wu G, Zhang L, Cheng Y, Hu C, Chen G, Zhang L, Liu X, Yan HH, Tan FL, Zhong W, Wu YL. Icotinib versus whole-brain irradiation in patients with EGFR-mutant non-small-cell lung cancer and multiple brain metastases (BRAIN): a multicentre, phase 3, open-label, parallel, randomised controlled trial. Lancet Respir Med. 2017 Sep;5(9):707-716. doi: 10.1016/S2213-2600(17)30262-X. Epub 2017 Jul 19. PMID 28734822
- [Background] Reungwetwattana T, Nakagawa K, Cho BC, Cobo M, Cho EK, Bertolini A, Bohnet S, Zhou C, Lee KH, Nogami N, Okamoto I, Leighl N, Hodge R, McKeown A, Brown AP, Rukazenkov Y, Ramalingam SS, Vansteenkiste J. CNS Response to Osimertinib Versus Standard Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors in Patients With Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Aug 28:JCO2018783118. doi: 10.1200/JCO.2018.78.3118. Online ahead of print. PMID 30153097
- [Derived] Yu Y, Pan Y, Zhou J, Mu S, Lu S. Dacomitinib in the treatment of EGFR-mutated non-small cell lung cancer with brain metastases: an open-label, multicenter, phase II study. Lung Cancer. 2025 Sep;207:108710. doi: 10.1016/j.lungcan.2025.108710. Epub 2025 Aug 11. PMID 40811939